CLINICAL TRIAL: NCT06203639
Title: Development and Preliminary Evaluation of an App to Reduce Caregiver Stress and Burden Among Informal Caregivers of People Living With Dementia
Brief Title: Evaluation of an App to Alleviate Stress Among Caregivers of People With Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-069
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Burden
Keywords: Dementia; mobile app
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the three group conditions: 1) UR Caregiver; 2) active control group; and 2) control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- UR Caregiver group (Experimental): Participants will be asked to use the UR Caregiver app daily (e.g., at least 15 minutes/day) for 8 weeks and complete and practice one module per week. On the eighth week, participants will be asked to review one of the past modules of their choice.
  Interventions: Other: UR Caregiver
- Active control (Active Comparator): Participants will be asked to use the app daily (e.g., at least 15 minutes/day) for an 8-week period.
  Interventions: Other: CLEAR Dementia Care
- Non-app using control (No Intervention): Participants in this group will not be using any apps in the study.

INTERVENTIONS:
Other: UR Caregiver — The UR Caregiver app was informed by previous research and developed in collaboration with caregiver partners. The app utilizes cognitive behavioural principles and is consistent with models of stress and coping. The app consists of seven modules. The app is available on IOS and Googe Play store. In addition to the didactic information provided in the app, worksheets are available in each module to practice the strategy/skill provided.
  Arms: UR Caregiver group
Other: CLEAR Dementia Care — A subset of participants will be randomly assigned to use the CLEAR Dementia Care app as part of an active control group. The app consists of features that primarily address care-related needs (as opposed to stress management strategies) allowing for a comparison with the UR Caregiver app. The app was developed by the Northern Health and Social Care Trust (Northern Ireland) and is freely available on both IOS and Google Play stores. The CLEAR Dementia Care app provides users with information about dementia (e.g., the different types of dementia, how dementia affects the brain, and symptoms associated with dementia). The app offers suggestions and alternative approaches to various care-related situations through illustrations/images that caregivers may experience.
  Arms: Active control

SUMMARY:
Caregivers of people living with dementia experience significant stress which can negatively affect their mental health. The goal of our study is to test a newly developed app that focuses on providing stress management strategies for caregivers of people living with dementia.

DETAILED DESCRIPTION:
Caregivers of people living with dementia experience significant stress which can negatively affect their mental health. Psychological interventions that focus on building skills and providing strategies to improve their well-being have been shown to improve caregiver well-being. Although mobile applications (apps) are available for caregivers of people living with dementia, existing apps do not adequately address the stress and mental health needs experienced by caregivers of people living with dementia. In addition, there is a paucity of mobile app interventions that provide practical stress management strategies for caregivers. The goal of the study is to conduct an evaluation of a novel app (UR Caregiver) that focuses on providing stress management strategies for caregivers of people living with dementia. The app utilizes cognitive behavioural principles and is consistent with models of stress and coping. Caregivers of people living with dementia will be recruited and randomly assigned to three groups: 1) UR Caregiver; 2) active control; and 3) non-app using control. Participants in the app-using groups will be asked to use the app over an 8-week period. Stress, burden, and mental health will be assessed before, after the 8-week period, and at a follow-up period. A 3 between (group) by 3 within (time: baseline, post, follow-up) mixed model (repeated measures) multivariate analysis of variance and univariate analyses will be conducted to examine improvements on outcome measures over time. Given the demands that caregivers of people living with dementia face daily, the creation and evaluation of an app that aims to provide stress-management strategies has the potential of improving the quality of life of caregivers of people living with dementia.

ELIGIBILITY:
Inclusion Criteria:

1. caregivers providing informal and unpaid care (e.g., spouses, children, relatives) for a person living with dementia
2. providing primary care (i.e., most of the care or equally shares the care with another individual such as a mother or sibling) for the person living with dementia
3. own a smartphone/tablet (i.e., can access either IOS or Android platforms).

Exclusion Criteria:

1) Currently using an app for caregiver stress/burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Perceived Stress Scale-10 (PSS-10) total scores at 8-weeks | The PSS-10 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload over the past month. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress
Change from baseline in the Perceived Stress Scale-10 (PSS-10) total scores at a 4-week follow-up | The PSS-10 will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow-up period
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload over the past month. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress
Change from after the 8-week period in the Perceived Stress Scale-10 (PSS-10) total scores at a 4-week follow-up | The PSS-10 will be administered immediately after the 8-week period and at a 4-week follow-up period
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload over the past month. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress
Change from baseline in the Burden Scale for Family Caregivers-Short Version (BSFC-S) total scores at 8-weeks | The BSFC-S will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  Subjective caregiver burden will be assessed using the BSFC-S. The BSFC-S is a 10-item scale developed to assess subjective burden. The BSFC-S was derived from the original 28-item scale. Each item is rated on a scale from 0 (Strongly disagree) to 3 (Strongly agree). Responses are summed with total scores ranging from 0 to 30 points with higher scores indicating greater caregiver burden
Change from baseline in the BSFC-S total scores at a 4-week follow-up | The BSFC-S will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow up
  Subjective caregiver burden will be assessed using the BSFC-S. The BSFC-S is a 10-item scale developed to assess subjective burden. The BSFC-S was derived from the original 28-item scale. Each item is rated on a scale from 0 (Strongly disagree) to 3 (Strongly agree). Responses are summed with total scores ranging from 0 to 30 points with higher scores indicating greater caregiver burden
Change from after the 8-week period in the BSFC-S total scores at a 4-week follow-up | The BSFC-S will be administered immediately after the 8-week period and at a 4-week follow-up period
  Subjective caregiver burden will be assessed using the BSFC-S. The BSFC-S is a 10-item scale developed to assess subjective burden. The BSFC-S was derived from the original 28-item scale. Each item is rated on a scale from 0 (Strongly disagree) to 3 (Strongly agree). Responses are summed with total scores ranging from 0 to 30 points with higher scores indicating greater caregiver burden
Change from baseline in the Patient Health Questionnaire-9 (PHQ-9) total scores at 8-weeks | The PHQ-9 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  The PHQ-9 is a 9-item self-report instrument widely used to assess for the presence and frequency of depressive symptoms over the last two weeks. Each of the nine items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 27) is calculated with increasing scores indicating greater depressive symptoms.
Change from baseline in the PHQ-9 total scores at a 4-week follow-up | The PHQ-9 will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow-up period
  The PHQ-9 is a 9-item self-report instrument widely used to assess for the presence and frequency of depressive symptoms over the last two weeks. Each of the nine items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 27) is calculated with increasing scores indicating greater depressive symptoms.
Change from after the 8-week period in the PHQ-9 total scores at a 4-week follow-up | The PHQ-9 will be administered immediately after the 8-week period and at a 4-week follow-up period
  The PHQ-9 is a 9-item self-report instrument widely used to assess for the presence and frequency of depressive symptoms over the last two weeks. Each of the nine items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 27) is calculated with increasing scores indicating greater depressive symptoms.
Change from baseline in the Generalized Anxiety Disorder-7 (GAD-7) total scores at 8-weeks | The GAD-7 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  The GAD-7 is a 7-item self-report instrument widely used to assess for anxiety symptoms. Each of the seven items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 21) is calculated with increasing scores indicating greater anxiety symptoms.
Change from baseline in the GAD-7 total scores at a 4-week follow-up | The GAD-7 will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow up period
  The GAD-7 is a 7-item self-report instrument widely used to assess for anxiety symptoms. Each of the seven items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 21) is calculated with increasing scores indicating greater anxiety symptoms.
Change from after the 8-week period in the GAD-7 total scores at a 4-week follow-up | The GAD-7 will be administered immediately after the 8-week period and at a 4-week follow-up period
  The GAD-7 is a 7-item self-report instrument widely used to assess for anxiety symptoms. Each of the seven items is rated on a Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). A total score (e.g., from 0 to 21) is calculated with increasing scores indicating greater anxiety symptoms.

SECONDARY OUTCOMES:
Change from baseline in the Multidimensional Scale for Perceived Social Support (MSPSS) total scores at 8-weeks | The MSPSS will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  The MSPSS is a 12-item self-report scale that measures perceived social support across three areas (e.g., family, friends and significant others. Each item is rated on a 7-point Likert scale with responses ranging from 1 (very strongly disagree) to 7 (very strongly agree). Item ratings are summed with total scores ranging from 12-84 and higher scores indicating greater perceived support.
Change from baseline in the MSPSS total scores at a 4-week follow-up | The MSPSS will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow up period
  The MSPSS is a 12-item self-report scale that measures perceived social support across three areas (e.g., family, friends and significant others. Each item is rated on a 7-point Likert scale with responses ranging from 1 (very strongly disagree) to 7 (very strongly agree). Item ratings are summed with total scores ranging from 12-84 and higher scores indicating greater perceived support.
Change from after the 8-week period in the MSPSS total scores at a 4-week follow-up | The MSPSS will be administered immediately after the 8-week period and at a 4-week follow-up period
  The MSPSS is a 12-item self-report scale that measures perceived social support across three areas (e.g., family, friends and significant others. Each item is rated on a 7-point Likert scale with responses ranging from 1 (very strongly disagree) to 7 (very strongly agree). Item ratings are summed with total scores ranging from 12-84 and higher scores indicating greater perceived support.
Change from baseline in the Caregiving Self-Efficacy Scale (CSES-8) total scores at 8-weeks | The CSES-8 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  The CSES-8 is an 8-item self-report measure that measures caregiver self-efficacy. Respondents are asked to indicate their level of confidence in response to each item from 1 (not at all confident) to 10 (totally confident). Accordingly, a single score is calculated by averaging the responses for the items (i.e., possible scores range from 1-10) with higher mean scores indicating higher self-efficacy.
Change from baseline in the CSES-8 total scores at a 4-week follow-up | The CSES-8 will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow up period
  The CSES-8 is an 8-item self-report measure that measures caregiver self-efficacy. Respondents are asked to indicate their level of confidence in response to each item from 1 (not at all confident) to 10 (totally confident). Accordingly, a single score is calculated by averaging the responses for the items (i.e., possible scores range from 1-10) with higher mean scores indicating higher self-efficacy.
Change from after the 8-week period in the CSES-8 total scores at a 4-week follow-up | The CSES-8 will be administered immediately after the 8-week period and at a 4-week follow-up period
  The CSES-8 is an 8-item self-report measure that measures caregiver self-efficacy. Respondents are asked to indicate their level of confidence in response to each item from 1 (not at all confident) to 10 (totally confident). Accordingly, a single score is calculated by averaging the responses for the items (i.e., possible scores range from 1-10) with higher mean scores indicating higher self-efficacy.
Change from baseline in the Brief-Coping Orientation to Problems Experienced Inventory (Brief-COPE) subscale scores at 8-weeks | The Brief-COPE will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 8-week period)
  Brief-COPE is a 28-item measure developed to assess different coping strategies used by individuals in response to stress. Three subscales can be obtained accordingly: emotion-focused, problem-focused, and dysfunctional subscale.
Change from baseline in the Brief-COPE subscale scores at a 4-week follow-up | The Brief-COPE will be administered at baseline (i.e., prior to starting the study) and at a 4-week follow up period
  Brief-COPE is a 28-item measure developed to assess different coping strategies used by individuals in response to stress. Three subscales can be obtained accordingly: emotion-focused, problem-focused, and dysfunctional subscale.
Change from after the 8-week period in the Brief-COPE subscale scores at a 4-week follow-up | The Brief-COPE will be administered immediately after the 8-week period and at a 4-week follow-up period
  Brief-COPE is a 28-item measure developed to assess different coping strategies used by individuals in response to stress. Three subscales can be obtained accordingly: emotion-focused, problem-focused, and dysfunctional subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Non-identified numeric data will be made available to other researchers, following the publication of the results, upon reasonable request for a period of at least 7 years. Textual data from the interviews will not be shared to protect participant anonymity.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available to other researchers, following the publication of the results, upon reasonable request for a period of at least 7 years.
Access Criteria: Requests by researchers who wish to access the data can be directed to Thomas.Hadjistavropoulos@uregina.ca

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Graessel E, Berth H, Lichte T, Grau H. Subjective caregiver burden: validity of the 10-item short version of the Burden Scale for Family Caregivers BSFC-s. BMC Geriatr. 2014 Feb 20;14:23. doi: 10.1186/1471-2318-14-23. PMID 24555474
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Ritter PL, Sheth K, Stewart AL, Gallagher-Thompson D, Lorig K. Development and Evaluation of the Eight-Item Caregiver Self-Efficacy Scale (CSES-8). Gerontologist. 2022 Mar 28;62(3):e140-e149. doi: 10.1093/geront/gnaa174. PMID 33146727